CLINICAL TRIAL: NCT05015166
Title: Study of an Internet-delivered Treatment Based on Experiential Dynamic Psychotherapy for Social Anxiety Disorder
Acronym: STePS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stockholm University (Other)
Responsible Party: Principal Investigator, Per Carlbring, Professor, Stockholm University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STePS
Record Dates: First submitted 2021-08-09; First posted 2021-08-20 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Social Anxiety Disorder
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Internet delivered self-help program with therapist support (Experimental): The intervention consists of 8 therapist-supported self-help modules delivered over 8 weeks on a secure online platform. Modules consist of texts and video followed by exercises which they send to their therapist and receive feedback within a few days.
  The treatment is based on principles from affect-focused psychodynamic psychotherapy.
  Interventions: Behavioral: Experimental: Internet delivered self-help program with therapist support
- Internet delivered self-help program without therapist support (Active Comparator): The intervention consists of 8 self-help modules delivered over 8 weeks on a secure online platform. Modules consist of texts and video followed by exercises which the participants are encouraged to try. The treatment is based on principles from affect-focused psychodynamic psychotherapy.
  Interventions: Behavioral: Internet delivered self-help program without therapist support
- Waitlist (No Intervention): Participants will receive no intervention for 8 weeks.

INTERVENTIONS:
Behavioral: Experimental: Internet delivered self-help program with therapist support — During 8 weeks of treatment participants are taught how emotional conflicts may underlie and perpetuate symptoms of social anxiety. They are also taught how to observe their own anxiety and emotional avoidance (i.e. defenses) and how to gradually approach previously warded off feelings. The final part of the program contains material on how one may express previously warded off emotions to improve important relationships. The treatment program consists of text, videos and a series of experiential exercises which a therapist gives feedback on.
  Arms: Internet delivered self-help program with therapist support
Behavioral: Internet delivered self-help program without therapist support — During 8 weeks of treatment participants are taught how emotional conflicts may underlie and perpetuate symptoms of social anxiety. They are also taught how to observe their own anxiety and emotional avoidance (i.e. defenses) and how to gradually approach previously warded off feelings. The final part of the program contains material on how one may express previously warded off emotions to improve important relationships. The treatment program consists of text, videos and a series of experiential exercises.
  Arms: Internet delivered self-help program without therapist support

SUMMARY:
The aim of this randomized, controlled study is to examine an internet delivered, self-help program for social anxiety based on psychodynamic therapy. The study will compare three conditions: the psychodynamic program with therapist support, without therapist support and a waitlist control.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Fulfill the DSM-5 criteria for social anxiety disorder (Score > 60 on the self-assessment instrument LSAS-SR)
* Have access to a computer/smartphone/tablet with internet connection
* Be able to read and write Swedish.

Exclusion Criteria:

* Suicidal (within the previous month, assessed with the self-assessment instrument C-SSRS)
* Partaking in psychological treatment
* Ongoing treatment with psychopharmacological drugs with dose adjustments within the nearest month or planned dose adjustments.

The following self-reported diagnoses are excluded:

* Autism spectrum disorder
* Serious depression (Score ≥ 20 on the PHQ9)
* Indications of psychosis or bipolar disorder (type 1 or 2).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2023-01-12 (Actual)

PRIMARY OUTCOMES:
Liebowitz Social Anxiety Scale, Self-Report, (LSAS-SR) | Change from baseline to post-treatment (8 week) and follow up (6, 12 and 24 months after treatment)
  The LSAS-SR features 48 items assessing social anxiety symptoms.

SECONDARY OUTCOMES:
Generalised Anxiety Disorder 7- item scale (GAD-7) | Change from baseline to post-treatment (8 week) and follow up (6, 12 and 24 months after treatment)
  The GAD-7 features seven items for assessing anxiety and screening for generalized anxiety disorder.
Patient Health Questionnaire 9-item scale (PHQ-9) | Change from baseline to post-treatment (8 week) and follow up (6, 12 and 24 months after treatment)
  The PHQ-9 features nine items for assessing depression in a clinical context and screening of depression in the general population
Brunnsviken Brief Quality of Life Scale (BBQ) | Change from baseline to post-treatment (8 week) and follow up (6, 12 and 24 months after treatment)
  The BBQ features 12 items concerning 6 areas of life rated on importance and satisfaction.

OTHER OUTCOMES:
The Personality Inventory for DSM Short Form (PID-5) | Baseline
  The PID-5 is a self-rated measure of personality-related problems featuring 25 items.
The Difficulties in Emotion Regulation Scale (DERS) | Change from baseline to post-treatment (8 week) and follow up (6, 12 and 24 months after treatment)
  Features 30 items assessing psychological strategies for handling emotional distress.
Self-Compassion Scale short-form (SCS-SF) | Change from baseline, week 3 and 6, to post-treatment (8 weeks) and follow up (6, 12 and 24 months after treatment)
  The SCS-SF features 12 items to record self-compassion towards yourself in difficult life situations.
Defense Mechanism Rating Scale, Self-Report-30 (DMRS-SR-30) | Change from baseline to post-treatment (8 week)
  DMRS-SR-30 features 30 items assessing psychological factors that influence emotional distress and quality of life.
Reflective Functioning Questionnaire 8 (RFQ-8) | Change from baseline, treatment week 1-8, to post-treatment (8 weeks).
  RFQ features 8 items assessing the ability to understand mental states of the self and others.
Internet Intervention Patient Adherence Scale | Change from baseline, and week 4, to post-treatment (8 weeks).
  iiPAS is rated by a clinician and features 5 items assessing a particular patient's adherence to internet-delivered psychological interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Per Carlbring, PhD, Principal Investigator — Department of Psychology at Stockholm University
Locations (1):
- Stockholm University, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Parts will be shared in an open data repository.

REFERENCES:
- [Derived] Mechler J, Lindqvist K, Magnusson K, Ringstrom A, Krafman JD, Alvinzi P, Kassius L, Sowa J, Andersson G, Carlbring P. Guided and unguided internet-delivered psychodynamic therapy for social anxiety disorder: A randomized controlled trial. Npj Ment Health Res. 2024 May 10;3(1):21. doi: 10.1038/s44184-024-00063-0. PMID 38730030